CLINICAL TRIAL: NCT04264546
Title: A Phase Ib Study to Evaluate the Safety and Immunogenicity of a Sabin Inactivated Poliovirus Vaccine (Vero Cell)
Brief Title: Safety and Immunogenicity of a Sabin Inactivated Poliovirus Vaccine (Phase Ib)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017L00935-1
Record Dates: First submitted 2020-02-09; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Polio
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Adult Group - High dosage (Experimental): One intramuscular injection of the investigational vaccine (0.5 ml); Intervention: one-dose regimen of high dosage investigational sIPV Intervention: Biological: one-dose regimen of high dosage investigational sIPV
  Interventions: Biological: sIPV
- Experimental Children Group - High dosage (Experimental): One intramuscular injection of the investigational vaccine (0.5 ml); Intervention: one-dose regimen of high dosage investigational sIPV Intervention: Biological: one-dose regimen of high dosage investigational sIPV
  Interventions: Biological: sIPV
- Experimental Infant Group - High dosage (Experimental): Three intramuscular injections of the investigational vaccine (0.5 ml) on Day 0, Day 30 and Day 60 respectively; Intervention: Three-dose regimen of high dosage investigational sIPV Intervention: Biological: Three-dose regimen of high dosage investigational sIPV
  Interventions: Biological: sIPV

INTERVENTIONS:
Biological: sIPV — The investigational High dosage Sabin IPV was all developed by Minhai Biotech Co., LTD. The antigen contents of type I, type II and type III polioviruses in the high dosage Sabin IPV were 22 DU, 65 DU and 65 DU. The vaccine was in liquid form, 0.5 ml per dose.

SUMMARY:
The purpose of this phase Ib study is to evaluate the safety of a Sabin Inactivated Poliovirus Vaccine (sIPV) in adults and children, and the safety and immunogenicity of it in infants. 20 adults aged 18~45 years and 20 children aged 4 years were only administered one dose of sIPV with high D antigen content. 20 infants aged 2 months (60~90 days) were administered three doses of sIPV with high D antigen content, on the month 0, 1, 2 schedule. Serum samples were collected before the 1st dose and 30 days after the 3rd dose vaccination to assess the immunogenicity in infants. Adverse events occurring within 30 days after each dose were collected to assess the safety.

DETAILED DESCRIPTION:
The purpose of this phase Ib study is to evaluate the safety of a Sabin Inactivated Poliovirus Vaccine (sIPV) in adults and children, and the safety and immunogenicity of it in infants. 20 adults aged 18~45 years and 20 children aged 4 years were only administered one dose of sIPV with high D antigen content. 20 infants aged 2 months (60~90 days) were administered three doses of sIPV with high D antigen content, on the month 0, 1, 2 schedule. Serum samples were collected before the 1st dose and 30 days after the 3rd dose vaccination to assess the immunogenicity in infants. Adverse events occurring within 30 days after each dose were collected to assess the safety.

The antigen contents of type I, type II and type III polioviruses in the high-dose Sabin IPV were 22 DU, 65 DU and 65 DU. All vaccines were in liquid form, 0.5 ml per dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer aged 18~45 years with/without prior vaccination of poliovirus and without any contraindication for vaccination;
* Healthy volunteer aged 4 years with/without prior vaccination of poliovirus but without booster vaccination and any contraindication for vaccination;
* Healthy volunteer aged 2 months (60~90 days) without prior vaccination of poliovirus and any contraindication for vaccination;
* Guardians of the participants should be capable of understanding the written consent form, and such form should be signed prior to enrolment;
* Complying with the requirement of the study protocol;
* Axillary temperature ≤ 37.0 °C;

Exclusion Criteria:

* Women aged 18~45 years with positive urine pregnancy test, pregnant or lactating women, or women with pregnancy plans within 3 months;
* Preterm or low birth weight infants;
* Congenital malformation, developmental disorders, genetic defects, or severe malnutrition;
* History of polio;
* Severe nervous system disease (epilepsy, seizures or convulsions) or mental illness;
* History of allergy to any vaccine, or any ingredient of the vaccine, or serious adverse reaction(s) to vaccination, such as urticaria, dyspnea, angioneurotic edema, abdominal pain, etc;
* Autoimmune disease or immunodeficiency/immunosuppressive;
* Bleeding disorder diagnosed by a doctor (e.g., coagulation factor deficiency, coagulation disorder, or platelet disorder), or significant bruising or coagulopathy;
* Serious chronic diseases, respiratory diseases, cardiovascular diseases, liver or kidney diseases or skin diseases;
* Mother of the participant has HIV infection;
* Acute illness or acute exacerbation of chronic disease within the past 7 days;
* Had a high fever within the past 3 days (axillary temperature ≥ 38.0°C);
* Receipt of any subunit or inactivated vaccine within the past 7 day;
* Receipt of any live attenuated vaccine within the past 14 days;
* Receipt of any blood product within the past 3 months;
* Any other factor that, in the judgment of the investigator, suggesting the volunteer is unsuitable for this study;

Ages: 60 Days to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
The seroconversion rates (SCRs) of each group 30 days after three-dose regimen | 28~42 days
  Subjects whose pre-immune antibody level < 1:8 and post-immune antibody level ≥ 1:8, or those whose pre-immune antibody level ≥ 1:8 and the increase of post-immune antibody level ≥ 4 folds are considered seroconverted.
The geometric mean titer (GMT) of each group 30 days after three-dose regimen | 28~42 days
  GMT of each group 28~42 days after three-dose regimen
The geometric mean fold increase (GMI) of each group 30 days after three-dose regimen | 28~42 days
  The GMI is the increase of post-immune GMT from pre-immune GMT

SECONDARY OUTCOMES:
The incidences of adverse reactions of each group occurred within 30 days after each injection | 30 days
  The number of participants who had adverse reactions divided by the number of all participants
The incidences of adverse events (AEs) of each group occurred within 30 days after each injection | 30 days
  The number of participants who had adverse events (AEs) divided by the number of all participants

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, Master, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Disease Control and Prevention, Nanjing, China

REFERENCES:
- [Derived] Jia S, Tang R, Li G, Hu Y, Liang Q. The effect of maternal poliovirus antibodies on the immune responses of infants to poliovirus vaccines. BMC Infect Dis. 2020 Aug 31;20(1):641. doi: 10.1186/s12879-020-05348-1. PMID 32867698